CLINICAL TRIAL: NCT07052123
Title: Non-Invasive Blood Pressure Monitoring in ICU Patients Using the DARE Device
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier de Saint-Denis (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 0060_DARE
Record Dates: First submitted 2025-06-05; First posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Hemodynamics; Blood Pressure Monitoring; Intensive Care Units; Critical Illness; Monitoring, Physiologic
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MultiSense® Non-Invasive Hemodynamic Monitoring Arm (Experimental)
  Interventions: Device: MultiSense® Non-Invasive Hemodynamic Monitoring Device

INTERVENTIONS:
Device: MultiSense® Non-Invasive Hemodynamic Monitoring Device — The MultiSense® device is a wireless, non-invasive monitoring system designed to continuously measure blood pressure, microcirculation, central body temperature, and detect arrhythmias in ICU patients. It aims to reduce risks associated with invasive monitoring, improve patient comfort and mobility, and decrease alarm fatigue through intelligent alert algorithms.

SUMMARY:
This study tests a new non-invasive device called DARE to monitor blood pressure in patients in intensive care. It compares the device's readings to standard invasive methods and also looks at how well it measures other vital signs like temperature, oxygen levels, and heart rhythm. The goal is to improve patient safety and comfort while helping doctors detect problems earlier.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (male or female), aged 18 years or older
* Admitted to intensive care unit (ICU) or critical care with an expected hospital stay longer than 2 days
* Equipped with an arterial catheter for invasive blood pressure monitoring
* Equipped with a urinary catheter for invasive core body temperature monitoring

Exclusion Criteria:

* Patients under 18 years old (minors)
* Known skin allergy to adhesives or silicone, or skin condition preventing adhesive use
* History of extensive skin pathology (e.g., Lyell syndrome)
* Patients with therapeutic limitations
* Patients with active implanted medical devices (e.g., pacemaker, defibrillator)
* Pregnant or breastfeeding women
* Patients not affiliated with the French social security system
* Patients or their legal representatives refusing consent, or unable to understand information and give informed consent
* Patients under legal guardianship, curatorship, or deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2025-03-24 (Actual); Primary Completion 2028-03-24 (Estimated); Study Completion 2028-03-24 (Estimated)

PRIMARY OUTCOMES:
Primary outcome: Agreement between non-invasive blood pressure index (IPA) from MultiSense® and invasive blood pressure (PAI) from ICU monitors. | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- France, Saint-Denis, France, France